CLINICAL TRIAL: NCT02514512
Title: Phase I Feasibility Study of Lung Cancer Radiotherapy Using Realtime Dynamic Multileaf Collimator (MLC) Adaptation and Radiofrequency Tracking
Brief Title: Lung Cancer Radiotherapy Using Realtime Dynamic Multileaf Collimator (MLC) Adaptation And Radiofrequency Tracking
Acronym: LIGHTSABR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Collaborators: University of Sydney (Other); Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC/15/HAWKE/55
Record Dates: First submitted 2015-07-12; First posted 2015-08-03 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms; Lung Neoplasms
Keywords: Lung Cancer; Stereotactic Ablative Radiotherapy (SABR); MLC Tracking; Radiotherapy
MeSH Terms: conditions — Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard SABR (No Intervention): Patients receive standard treatment
- MLC Tracking SABR (Experimental): Patients are treated with MLC tracking
  Interventions: Device: MLC Tracking

INTERVENTIONS:
Device: MLC Tracking — Treat patient with Non FDA approved MLC Tracking
  Arms: MLC Tracking SABR

SUMMARY:
A research study into a new technology for adjustment of the radiotherapy beam to account for movement of lung tumours as the patient breathes during radiotherapy.

DETAILED DESCRIPTION:
Twenty patients 18 years of age or more and undergoing Stereotactic Body Radiotherapy (SBRT) at Northern Sydney Cancer Centre for lung cancer will receive the new treatment. Participants will be physically able to undergo all aspects of treatment and intellectually able to provide written informed consent and complete questionnaires. Beacons will be implanted in the patients' lung to allow the Multi Leaf Collimator (MLC) tracking equipment to follow precisely the movement of the lung. The difference in ability to track tumour movement between MLC and the current standard method will be compared to identify changes in study outcomes. Audiovisual (AV) Biofeedback will also be used to regulate patients' breathing during radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Has provided written Informed Consent for participation in this trial and is willing to comply with the study
* Patients undergoing external beam radiotherapy at Northern Sydney Cancer Centre
* Histologically proven Stage I Non Small Cell Lung Cancer (NSCLC) oligometastatic lung metastases (3 or less). Histological diagnosis will be obtained if clinically indicated.
* MRI/4D-CT prior to insertion of Calypso beacons
* Patient must be able to have Varian Calypso beacons placed in the lung (if on anticoagulants, must be cleared by Local Medical Officer (LMO) or cardiologist).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Body habitus enabling Calypso tracking (as per Calypso Determining a Patient's Localisation Designation & Orientation before implantation)
* A maximum of three metastases to the lung from any non-haematological malignancy. Multiple metastases will be treated separately.
* Tumour diameter ≤ = 5cm

Exclusion Criteria:

* Previous high-dose thoracic radiotherapy.
* Less than two Calypso beacons implanted in the lung.
* Calypso beacons are spaced by greater than 9cm or less than 1cm.
* Calypso beacons are less than 19cm from outer chest wall
* Cytotoxic chemotherapy within 3 weeks of commencement of treatment, or concurrently with treatment. Hormonal manipulation agents are allowable (e.g. aromatase inhibitors, selective oestrogen receptor modulators, and gonadotropin releasing hormone receptor modulators)
* Targeted agents (such as sunitinib, bevacizumab and tarceva) within 7 days of commencement of treatment, or concurrently with treatment
* Women who are pregnant or lactating.
* Unwilling or unable to give informed consent
* Unwilling or unable to complete quality of life questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To demonstrate feasibility of MLC tracking for lung cancer | Assessed at 2 years
  Percentage of fractions delivered without software or mechanical failure

SECONDARY OUTCOMES:
Audio Visual (AV) Biofeedback | Assessed at 2 years
  Fraction of patients for whom AV biofeedback improves breathing regularity
Coefficient of variation in breathing patterns | Assessed at 2 years
  Breathing variations over imaging and treatment sessions with and without AV biofeedback using a statistical process for coefficient of variation
Target volumes | Assessed at 2 years
  Target volumes between the 4 Dimensional (4D) planning MLC tracking and Internal Target Volume (ITV) (standard) planning
Lung dose | Assessed at 2 years
  Difference in dose to healthy lung in treatment plans between 4D planning and ITV planning
Treated dose - MLC tracking | Assessed at 2 years
  Difference between the treated dose and planned dose for MLC tracking
Treated dose - standard | Assessed at 2 years
  Difference between the estimated treated dose and planned dose for ITV treatments
4D Cone Beam CT (CBCT) image quality | Assessed at 2 years
  Image quality and target position differences between the Calypso-based 4D CBCT image reconstruction and Revs Per Minute (RPM)-based 4D CBCT image reconstruction using Feldkamp filtered backprojection (FDK and iterative reconstruction algorithms.
Breathing variations with and without continuous positive air pressure (CPAP) | At time of treatment
  To quantify the breathing variations over treatment sessions with and without application of continuous positive air pressure (CPAP)

OTHER OUTCOMES:
Patient Outcomes - Composite | 5 years
  Participants will be followed for 5 years to determine patient outcome3s, including radiation therapy toxicity, local control (whether the tumour has spread) and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eade, MD, Principal Investigator — RNSH
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data is to be shared with USyd to fulfil the secondary endpoints of the trial

REFERENCES:
- [Derived] Caillet V, Zwan B, Briggs A, Hardcastle N, Szymura K, Prodreka A, O'Brien R, Harris BE, Greer P, Haddad C, Jayamanne D, Eade T, Booth J, Keall P. Geometric uncertainty analysis of MLC tracking for lung SABR. Phys Med Biol. 2020 Dec 2;65(23):235040. doi: 10.1088/1361-6560/abb0c6. PMID 33263318
- [Derived] Booth J, Caillet V, Briggs A, Hardcastle N, Angelis G, Jayamanne D, Shepherd M, Podreka A, Szymura K, Nguyen DT, Poulsen P, O'Brien R, Harris B, Haddad C, Eade T, Keall P. MLC tracking for lung SABR is feasible, efficient and delivers high-precision target dose and lower normal tissue dose. Radiother Oncol. 2021 Feb;155:131-137. doi: 10.1016/j.radonc.2020.10.036. Epub 2020 Nov 3. PMID 33152399